CLINICAL TRIAL: NCT05932225
Title: Systane® Complete Preservative Free Lubricant Eye Drops
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEC262-I001
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Systane Complete Preservative-Free (Experimental): 1-2 drops in each eye four times a day for 30 days
  Interventions: Other: Propylene glycol solution/drops

INTERVENTIONS:
Other: Propylene glycol solution/drops — Commercially available eye drops
  Other Names: Systane Complete Preservative-Free

SUMMARY:
The purpose of this post-market clinical follow-up (PMCF) study is to assess the performance and safety of Systane Complete Preservative Free (PF) lubricant eye drops in subjects experiencing dry eye symptoms. Statistical analyses will be presented overall and by Dry Eye Disease (DED) group.

DETAILED DESCRIPTION:
Subjects will participate in the study for approximately 30 days, with a Screening/Baseline visit scheduled on Day 1, a phone call scheduled on Day 15 ± 2 (Visit 2) and a follow-up visit scheduled on Day 30 ± 2 (Visit 3). Subjects will be asked to complete the Impact of Dry Eye on Everyday Life - Symptom Bother [IDEEL-SB]) questionnaire on Day 1 and Visit 3. In addition, subjects will be instructed to document Systane Complete PF dosing information on a daily basis using a subject diary.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be able to understand and sign an informed consent form
* Subject with mild to moderate dry eye
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Has suffered any ocular injury to either eye in the past 3 months prior to screening.
* Has undergone any other ocular surgery (including intraocular surgery) within the past 6 months or has any ocular surgery planned during the study.
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (4):
- Canada (4):
  - Integra Eye Care, Burnaby, British Columbia
  - Aggarwal and Associates Limited, Brampton, Ontario
  - Eyes on Sheppard Clinic, North York, Ontario
  - University of Waterloo Centre for Contact Lens Research, Waterloo, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 4 investigative sites located in Canada.
Pre-assignment Details: Of the 71 enrolled, 3 participants did not meet the inclusion criteria and were exited from the study. This reporting group includes all eligible subjects (68).
Groups:
- Aqueous Deficient Dry Eye: 1-2 drops of Systane Complete PF in each eye four times a day for 30 days. Participants in this group experienced dry eye symptoms due to insufficient tear gland production.
- Evaporative Dry Eye: 1-2 drops of Systane Complete PF in each eye four times a day for 30 days. Participants in this group experienced dry eye symptoms due to insufficient oil in their tears (meibomian gland dysfunction).
- Mixed Dry Eye: 1-2 drops of Systane Complete PF in each eye four times a day for 30 days. Participants in this group experienced dry eye symptoms due to insufficient tear gland production and insufficient oil in their tears (meibomian gland dysfunction).
Period: Overall Study
Arm/Group | Aqueous Deficient Dry Eye | Evaporative Dry Eye | Mixed Dry Eye
Started | 14 | 32 | 22
Completed | 13 | 29 | 22
Not Completed | 1 | 3 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — As detailed in the Clinical Study Report | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All eligible participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Aqueous Deficient Dry Eye | Evaporative Dry Eye | Mixed Dry Eye | Total
Number analyzed (Participants) | 14 | 32 | 22 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (17.62) | 49.2 (14.34) | 55.0 (11.99) | 51.1 (14.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 24 | 11 | 47
  Male | 2 | 8 | 11 | 21
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 3 | 10 | 3 | 16
  Not Hispanic or Latino | 11 | 21 | 19 | 51
  Unknown | 0 | 1 | 0 | 1
  Unconfirmed | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 11 | 10 | 22
  Black or African American | 0 | 2 | 0 | 2
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0
  White | 8 | 9 | 9 | 26
  Mixed | 0 | 0 | 0 | 0
  Other | 1 | 1 | 1 | 3
  Unknown | 4 | 9 | 2 | 15
  Unconfirmed | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 14 | 32 | 22 | 68

OUTCOME MEASURES:

1. Primary Outcome: Mean Overall Impact of Dry Eye on Everyday Life Symptom Bother (IDEEL SB) Score - By Dry Eye Group
Description: The IDEEL SB module is a 20-question, patient-reported outcome questionnaire that assesses the subject's symptoms of dry eye. For each question, the subject selected a single response for both eyes, where 0="None of the time" (Q1) or "I did not have this symptom/Not Applicable" (Q2-20) to 4="All of the time" (Q1) or "Very Much" (Q2-20). The overall Symptom Bother score was calculated as the mean value of the non-missing item scores (Q1-20) multiplied by 25, for an overall resultant score ranging from 0 to 100. Higher scores indicate greater symptom bother. No statistical hypothesis was pre-specified for this endpoint.
Time Frame: Baseline (Day 1 pretreatment), Day 30
Population: Full Analysis Set: All subjects/eyes exposed to at least one dose of Systane Complete PF with data at visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aqueous Deficient Dry Eye | Evaporative Dry Eye | Mixed Dry Eye
Number analyzed (Participants) | 14 | 32 | 22
score on a scale
  Baseline (Day 1 pretreatment) | 41.36 (11.095) | 47.08 (12.689) | 47.63 (11.756)
  Day 30: number analyzed (Participants) | 13 | 29 | 22
  Day 30 | 31.26 (9.449) | 32.16 (11.080) | 32.91 (10.016)

2. Primary Outcome: Mean Overall Impact of Dry Eye on Everyday Life Symptom Bother (IDEEL SB) Score - All Subjects
Description: as for outcome 1
Time Frame: Baseline (Day 1 pretreatment), Day 30
Population: Full Analysis Set: All subjects/eyes exposed to at least one dose of Systane Complete PF with data at visit
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Systane Complete PF: 1-2 drops of Systane Complete PF in each eye four times a day for 30 days.
Arm/Group | Systane Complete PF
Number analyzed (Participants) | 68
score on a scale
  Baseline (Day 1 pretreatment) | 46.08 (12.150)
  Day 30: number analyzed (Participants) | 64
  Day 30 | 32.24 (10.265)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent until study exit. The total expected duration of participation for each subject was approximately 30 days.
Description: AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is included with unit of "eyes." The Other (Not Including Serious) Adverse Event table reports only the AEs that occurred above a 5% threshold in one or more reporting group. This analysis population includes all subjects/eyes exposed to at least one dose of Systane Complete PF.
Groups:
- Pretreatment: All subjects prior to exposure to Systane Complete PF
- Aqueous Deficient Dry Eye - Ocular; Aqueous Deficient Dry Eye - Nonocular; Evaporative Dry Eye - Ocular; Evaporative Dry Eye - Nonocular; Mixed Dry Eye - Ocular; Mixed Dry Eye - Nonocular: Subgroup of subjects exposed to at least one dose of Systane Complete PF
- Overall - Ocular; Overall - Nonocular: All subjects exposed to at least one dose of Systane Complete PF
Arm/Group | Pretreatment | Aqueous Deficient Dry Eye - Ocular | Aqueous Deficient Dry Eye - Nonocular | Evaporative Dry Eye - Ocular | Evaporative Dry Eye - Nonocular | Mixed Dry Eye - Ocular | Mixed Dry Eye - Nonocular | Overall - Ocular | Overall - Nonocular
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/28 | 0/14 | 0/64 | 0/32 | 0/44 | 0/22 | 0/136 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/28 | 0/14 | 0/64 | 0/32 | 0/44 | 0/22 | 0/136 | 0/68
Other Adverse Events (participants affected / at risk) | 0/68 | 0/28 | 0/14 | 0/64 | 0/32 | 0/44 | 0/22 | 0/136 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/25/NCT05932225/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/25/NCT05932225/SAP_001.pdf